CLINICAL TRIAL: NCT04758403
Title: Cone Beam Computed Tomography - Guided Navigation Bronchoscopy for Peripheral Pulmonary Nodules: A Randomized Trial
Brief Title: CBCT-Guided Navigational Bronchoscopy For Lung Nodules
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to changes in technology (EMN technology replaced by robotic platform) the study was terminated
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Philips Healthcare (Industry); Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Adnan Majid, MD, Principal Investigator, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 20-580
Record Dates: First submitted 2021-02-14; First posted 2021-02-17 (Actual); Results first posted 2024-11-19 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-10

CONDITIONS: Peripheral Pulmonary Nodules; Lung; Node; Cone Beam Computed Tomography; Guided Navigation Bronchoscopy
Keywords: Peripheral Pulmonary Nodules; Lung; Node; Cone Beam Computed Tomography; Guided Navigation Bronchoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Navigation Bronchoscopy ALONE (Experimental): This research study involves a screening period, a procedure and follow up visits
  * Procedure Visit Navigation Bronchoscopy Alone
  * Follow-Up Visits at Week 1, 4 and 12
  Interventions: Radiation: Navigation Bronchoscopy
- CBCT-GUIDED Navigation Bronchoscopy (Experimental): This research study involves a screening period, a procedure and follow up visits Procedure Visit- Cone Beam Computed Tomography - Guided Navigation Bronchoscopy for Peripheral Pulmonary Nodules
  -Follow-Up Visits at Week 1, 4 and 12
  Interventions: Radiation: Navigation Bronchoscopy; Radiation: Cone beam computed tomography (CBCT)

INTERVENTIONS:
Radiation: Navigation Bronchoscopy — Navigation Bronchoscopy procedure will be performed per product instructions and the institution's standard practice.
  Other Names: NB
Radiation: Cone beam computed tomography (CBCT) — Per Protocol
  Arms: CBCT-GUIDED Navigation Bronchoscopy

SUMMARY:
The purpose of this study is to determine if the cone beam computed tomography (CBCT)-guided navigation bronchoscopy is better in diagnosing lung nodules compared to navigation bronchoscopy alone.

DETAILED DESCRIPTION:
This clinical trial examines the effectiveness of a treatment comparing it to another known treatment.

The U.S. Food and Drug Administration (FDA) has approved the navigation bronchoscopy as a treatment option for this disease.

The U.S. Food and Drug Administration (FDA) has approved the Cone-Beam CT scan as a treatment option for this disease.

This research study involves a screening period, a procedure and follow up visits.

The names of the study interventions involved in this study are:

* Computed tomography (CBCT)-guided navigation bronchoscopy (CBCT-guided NB)
* Navigation bronchoscopy alone

Participants will receive the study procedure and will be followed for up to 6 months.

It is expected that about 136 people will take part in this research study.

ELIGIBILITY:
Inclusion Criteria:

* Participants ≥18 years old.
* Participants with lesions having an intermediate pre-test probability of malignancy (pCA, 0.05 to 0.65) as determined by Swensen-Mayo nodule risk calculator and in whom bronchoscopic biopsy was determined to be the next best treatment step by the treating pulmonologist.
* Participants with higher risk lesions (pCA > 0.65) in need of a diagnosis for nonsurgical treatment or prior to surgery.
* Participants are willing and able to provide informed consent.

Exclusion Criteria:

* The participant is pregnant as confirmed by urine or serum pregnancy testing.
* There is a predetermined plan to pursue stereotactic body radiation therapy (SBRT) in the event of a nondiagnostic study procedure in participant's with a nodule in the outer 1/3 lung zone (i.e. The participant would not go on for a CT guided TTNA).
* Lacked fitness according to physician judgement to undergo bronchoscopy.
* Contraindication for temporary interruption of the use of anticoagulant therapy.
* Uncontrolled or irreversible coagulopathy.
* Known allergy for lidocaine.
* Uncontrolled pulmonary hypertension.
* Recent (< 4 weeks) and/or uncontrolled cardiac disease.
* Compromised upper airway (eg concomitant head and neck cancer or central airway stenosis such that endobronchial access is considered unsafe).
* ASA classification ≥ 4.
* COVID-19 positive participant at the time of procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-03-05 (Actual); Primary Completion 2023-04-12 (Actual); Study Completion 2023-04-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adnan Majid, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconness Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Sponsor Investigator or designee. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Beth Israel Deaconess Medical Center Technology Ventures Office at tvo@bidmc.harvard.edu

REFERENCES:
- [Background] Choi JW, Park CM, Goo JM, Park YK, Sung W, Lee HJ, Lee SM, Ko JY, Shim MS. C-arm cone-beam CT-guided percutaneous transthoracic needle biopsy of small (</= 20 mm) lung nodules: diagnostic accuracy and complications in 161 patients. AJR Am J Roentgenol. 2012 Sep;199(3):W322-30. doi: 10.2214/AJR.11.7576. PMID 22915422
- [Background] Hur J, Lee HJ, Nam JE, Kim YJ, Kim TH, Choe KO, Choi BW. Diagnostic accuracy of CT fluoroscopy-guided needle aspiration biopsy of ground-glass opacity pulmonary lesions. AJR Am J Roentgenol. 2009 Mar;192(3):629-34. doi: 10.2214/AJR.08.1366. PMID 19234257
- [Background] Ohno Y, Hatabu H, Takenaka D, Higashino T, Watanabe H, Ohbayashi C, Sugimura K. CT-guided transthoracic needle aspiration biopsy of small (< or = 20 mm) solitary pulmonary nodules. AJR Am J Roentgenol. 2003 Jun;180(6):1665-9. doi: 10.2214/ajr.180.6.1801665. PMID 12760939
- [Background] Laspas F, Roussakis A, Efthimiadou R, Papaioannou D, Papadopoulos S, Andreou J. Percutaneous CT-guided fine-needle aspiration of pulmonary lesions: Results and complications in 409 patients. J Med Imaging Radiat Oncol. 2008 Oct;52(5):458-62. doi: 10.1111/j.1440-1673.2008.01990.x. PMID 19032391
- [Background] DiBardino DM, Yarmus LB, Semaan RW. Transthoracic needle biopsy of the lung. J Thorac Dis. 2015 Dec;7(Suppl 4):S304-16. doi: 10.3978/j.issn.2072-1439.2015.12.16. PMID 26807279
- [Background] Wiener RS, Schwartz LM, Woloshin S, Welch HG. Population-based risk for complications after transthoracic needle lung biopsy of a pulmonary nodule: an analysis of discharge records. Ann Intern Med. 2011 Aug 2;155(3):137-44. doi: 10.7326/0003-4819-155-3-201108020-00003. PMID 21810706
- [Background] Ost DE, Ernst A, Lei X, Kovitz KL, Benzaquen S, Diaz-Mendoza J, Greenhill S, Toth J, Feller-Kopman D, Puchalski J, Baram D, Karunakara R, Jimenez CA, Filner JJ, Morice RC, Eapen GA, Michaud GC, Estrada-Y-Martin RM, Rafeq S, Grosu HB, Ray C, Gilbert CR, Yarmus LB, Simoff M; AQuIRE Bronchoscopy Registry. Diagnostic Yield and Complications of Bronchoscopy for Peripheral Lung Lesions. Results of the AQuIRE Registry. Am J Respir Crit Care Med. 2016 Jan 1;193(1):68-77. doi: 10.1164/rccm.201507-1332OC. PMID 26367186
- [Background] Ernst A, Simoff M, Ost D, Michaud G, Chandra D, Herth FJ. A multicenter, prospective, advanced diagnostic bronchoscopy outcomes registry. Chest. 2010 Jul;138(1):165-70. doi: 10.1378/chest.09-2457. Epub 2010 Apr 2. PMID 20363846
- [Background] Asano F, Aoe M, Ohsaki Y, Okada Y, Sasada S, Sato S, Suzuki E, Senba H, Fujino S, Ohmori K. Deaths and complications associated with respiratory endoscopy: a survey by the Japan Society for Respiratory Endoscopy in 2010. Respirology. 2012 Apr;17(3):478-85. doi: 10.1111/j.1440-1843.2011.02123.x. PMID 22222022
- [Background] Khandhar SJ, Bowling MR, Flandes J, Gildea TR, Hood KL, Krimsky WS, Minnich DJ, Murgu SD, Pritchett M, Toloza EM, Wahidi MM, Wolvers JJ, Folch EE; NAVIGATE Study Investigators. Electromagnetic navigation bronchoscopy to access lung lesions in 1,000 subjects: first results of the prospective, multicenter NAVIGATE study. BMC Pulm Med. 2017 Apr 11;17(1):59. doi: 10.1186/s12890-017-0403-9. PMID 28399830
- [Background] Ali EAA, Takizawa H, Kawakita N, Sawada T, Tsuboi M, Toba H, Takashima M, Matsumoto D, Yoshida M, Kawakami Y, Kondo K, Khairy El-Badrawy M, Tangoku A. Transbronchial Biopsy Using an Ultrathin Bronchoscope Guided by Cone-Beam Computed Tomography and Virtual Bronchoscopic Navigation in the Diagnosis of Pulmonary Nodules. Respiration. 2019;98(4):321-328. doi: 10.1159/000500228. Epub 2019 May 23. PMID 31121593
- [Background] Rivera MP, Mehta AC, Wahidi MM. Establishing the diagnosis of lung cancer: Diagnosis and management of lung cancer, 3rd ed: American College of Chest Physicians evidence-based clinical practice guidelines. Chest. 2013 May;143(5 Suppl):e142S-e165S. doi: 10.1378/chest.12-2353. PMID 23649436
- [Background] Mondoni M, Sotgiu G, Bonifazi M, Dore S, Parazzini EM, Carlucci P, Gasparini S, Centanni S. Transbronchial needle aspiration in peripheral pulmonary lesions: a systematic review and meta-analysis. Eur Respir J. 2016 Jul;48(1):196-204. doi: 10.1183/13993003.00051-2016. Epub 2016 May 12. PMID 27174878
- [Background] Pritchett MA, Schampaert S, de Groot JAH, Schirmer CC, van der Bom I. Cone-Beam CT With Augmented Fluoroscopy Combined With Electromagnetic Navigation Bronchoscopy for Biopsy of Pulmonary Nodules. J Bronchology Interv Pulmonol. 2018 Oct;25(4):274-282. doi: 10.1097/LBR.0000000000000536. PMID 30179922
- [Background] Gould MK, Donington J, Lynch WR, Mazzone PJ, Midthun DE, Naidich DP, Wiener RS. Evaluation of individuals with pulmonary nodules: when is it lung cancer? Diagnosis and management of lung cancer, 3rd ed: American College of Chest Physicians evidence-based clinical practice guidelines. Chest. 2013 May;143(5 Suppl):e93S-e120S. doi: 10.1378/chest.12-2351. PMID 23649456
- [Background] National Lung Screening Trial Research Team; Aberle DR, Adams AM, Berg CD, Black WC, Clapp JD, Fagerstrom RM, Gareen IF, Gatsonis C, Marcus PM, Sicks JD. Reduced lung-cancer mortality with low-dose computed tomographic screening. N Engl J Med. 2011 Aug 4;365(5):395-409. doi: 10.1056/NEJMoa1102873. Epub 2011 Jun 29. PMID 21714641
- [Background] Wang Memoli JS, Nietert PJ, Silvestri GA. Meta-analysis of guided bronchoscopy for the evaluation of the pulmonary nodule. Chest. 2012 Aug;142(2):385-393. doi: 10.1378/chest.11-1764. PMID 21980059
- [Background] Bowling MR, Brown C, Anciano CJ. Feasibility and Safety of the Transbronchial Access Tool for Peripheral Pulmonary Nodule and Mass. Ann Thorac Surg. 2017 Aug;104(2):443-449. doi: 10.1016/j.athoracsur.2017.02.035. Epub 2017 May 17. PMID 28527967
- [Background] Casal RF, Sarkiss M, Jones AK, Stewart J, Tam A, Grosu HB, Ost DE, Jimenez CA, Eapen GA. Cone beam computed tomography-guided thin/ultrathin bronchoscopy for diagnosis of peripheral lung nodules: a prospective pilot study. J Thorac Dis. 2018 Dec;10(12):6950-6959. doi: 10.21037/jtd.2018.11.21. PMID 30746241
- [Background] Eberhardt R, Anantham D, Herth F, Feller-Kopman D, Ernst A. Electromagnetic navigation diagnostic bronchoscopy in peripheral lung lesions. Chest. 2007 Jun;131(6):1800-5. doi: 10.1378/chest.06-3016. Epub 2007 Mar 30. PMID 17400670
- [Background] Popovich J Jr, Kvale PA, Eichenhorn MS, Radke JR, Ohorodnik JM, Fine G. Diagnostic accuracy of multiple biopsies from flexible fiberoptic bronchoscopy. A comparison of central versus peripheral carcinoma. Am Rev Respir Dis. 1982 May;125(5):521-3. doi: 10.1164/arrd.1982.125.5.521. PMID 7081810
- [Background] Shure D, Astarita RW. Bronchogenic carcinoma presenting as an endobronchial mass. Chest. 1983 Jun;83(6):865-7. doi: 10.1378/chest.83.6.865. PMID 6303712
- [Background] Chopra SK, Genovesi MG, Simmons DH, Gothe B. Fiberoptic bronchoscopy in the diagnosis of lung cancer comparison of pre-and post-bronchoscopy sputa, washings, bruchings and biopsies. Acta Cytol. 1977 Jul-Aug;21(4):524-7. PMID 269602
- [Background] Hohenforst-Schmidt W, Zarogoulidis P, Vogl T, Turner JF, Browning R, Linsmeier B, Huang H, Li Q, Darwiche K, Freitag L, Simoff M, Kioumis I, Zarogoulidis K, Brachmann J. Cone Beam Computertomography (CBCT) in Interventional Chest Medicine - High Feasibility for Endobronchial Realtime Navigation. J Cancer. 2014 Mar 9;5(3):231-41. doi: 10.7150/jca.8834. eCollection 2014. PMID 24665347
- [Background] Wallis S. Z-squared: The Origin and Application of χ 2. J Quant Linguist [Internet]. 2013 Nov 12 [cited 2020 Nov 4];20(4):350-78. Available from: http://www.tandfonline.com/doi/abs/10.1080/09296174.2013.830554

RESULTS

PARTICIPANT FLOW:
Groups:
- CBCT-GUIDED Navigation Bronchoscopy: This research study involves a screening period, a procedure and follow up visits Procedure Visit- Cone Beam Computed Tomography - Guided Navigation Bronchoscopy for Peripheral Pulmonary Nodules
  -Follow-Up Visits at Week 1, 4 and 12
  Navigation Bronchoscopy: Navigation Bronchoscopy procedure will be performed per product instructions and the institution's standard practice.
  Cone beam computed tomography (CBCT): Per Protocol
- Navigation Bronchoscopy ALONE: Patients undergoing navigational bronchoscopy alone (not with CBCT) for peripheral pulmonary nodules.
Period: Overall Study
Arm/Group | CBCT-GUIDED Navigation Bronchoscopy | Navigation Bronchoscopy ALONE
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Navigation Bronchoscopy ALONE: This research study involves a screening period, a procedure and follow up visits
  * Procedure Visit Navigation Bronchoscopy Alone
  * Follow-Up Visits at Week 1, 4 and 12
  Navigation Bronchoscopy: Navigation Bronchoscopy procedure will be performed per product instructions and the institution's standard practice.
- Total: Total of all reporting groups
Arm/Group | Navigation Bronchoscopy ALONE | CBCT-GUIDED Navigation Bronchoscopy | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 76 [69 to 80] | 79 [73 to 81] | 78 [72.5 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 6 | 7 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 9 | 8 | 17
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Overall Diagnostic Yield
Description: The overall diagnostic yield will be calculated by adding the number of true positives (TP) for both malignancy and benign disease in the numerator and dividing by the total number of procedures performed for each arm of the study.
  Proportions will be compared with the Chi-Square Test as this test is equivalent to the z-test of two proportions (26). A p-value <0.05 will be considered as statistically significant.
Time Frame: 6 months
Population: Enrolled before trial termination but no data were collected.
Arm/Group | Navigation Bronchoscopy ALONE | CBCT-GUIDED Navigation Bronchoscopy
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Overall Incidence of Procedure-related Complications
Description: To compare complications between navigational bronchoscopy alone and CBCT guided bronchoscopy.
Time Frame: 6 months
Population: Enrolled before trial termination but no data were collected.
Arm/Group | Navigation Bronchoscopy ALONE | CBCT-GUIDED Navigation Bronchoscopy
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Additional Diagnostic Procedures in Navigational Bronchoscopy Alone and CBCT Guided Bronchoscopy.
Description: To compare the need of additional diagnostic procedures in navigational bronchoscopy alone and CBCT guided bronchoscopy.
Time Frame: 6 Months
Population: Enrolled before trial termination but no data were collected.
Arm/Group | Navigation Bronchoscopy ALONE | CBCT-GUIDED Navigation Bronchoscopy
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Navigational Time in Bronchoscopy Alone and CBCT Guided Bronchoscopy.
Description: To compare the navigational time defined as the time between the start of catheter driving after registration until catheter is parked for biopsy.
Time Frame: 6 Months
Population: Enrolled before trial termination but no data were collected.
Arm/Group | Navigation Bronchoscopy ALONE | CBCT-GUIDED Navigation Bronchoscopy
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Navigation Bronchoscopy ALONE | CBCT-GUIDED Navigation Bronchoscopy
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-05-12): https://cdn.clinicaltrials.gov/large-docs/03/NCT04758403/Prot_SAP_000.pdf
  • Informed Consent Form (2020-01-31): https://cdn.clinicaltrials.gov/large-docs/03/NCT04758403/ICF_001.pdf